CLINICAL TRIAL: NCT04659993
Title: Cancer Within a Pandemic: A Telemental Health Intervention Designed to Augment Psychological Resilience Amidst Dual Health Threats
Brief Title: Cancer Within a Pandemic: A Telemental Health Intervention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accruals
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00070150; WFBCCC01520 (Other: Wake Forest Baptist Comprehensive Cancer Center); P30CA012197 (NIH)
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Results first posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Cancer; Survivorship; Depression, Anxiety
Keywords: Telemental intervention
MeSH Terms: conditions — Neoplasms; Depression; Anxiety Disorders | interventions — Self-Help Groups; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telemental Group (Experimental): The virtual group will be conducted within a secure platform such as Microsoft WebEx. Assessments (pre-, post-, mid-way) will be distributed through REDCap, a secure virtual platform, as will session handouts and forms.
  Interventions: Behavioral: Telemental Health Sessions, Support Groups and Questionnaires

INTERVENTIONS:
Behavioral: Telemental Health Sessions, Support Groups and Questionnaires — Participants will complete initial online questionnaires lasting about 25-30 minutes as well as attend weekly support group meetings online. After 4 weeks, participants will complete seven online follow-up questionnaires that should take no longer than 30 minutes and again at the end of the study.

SUMMARY:
The purpose of this research study is to test an online support group designed to help young adults who have had cancer treatment to manage their mood during a pandemic. Investigators hope to learn more about what effects a support group may have upon the health and well-being of young adults who have undergone cancer treatment by offering an online support group that teaches healthy coping skills in a practical and acceptable way. Investigators would also like to know if certain parts of the online material is more effective in helping subjects manage their mood.

DETAILED DESCRIPTION:
Primary Objective: To improve self-efficacy for young adult cancer survivors navigating pandemic conditions.

Secondary Objective: To reduce depression and anxiety levels through meaning-making.

ELIGIBILITY:
Inclusion Criteria:

* Documented cancer diagnosis within the Wake Forest Baptist Medical Center medical record;
* Outpatient Cancer Survivor (diagnosis, treatment, or post-treatment);
* Aged 18-39
* Must speak English
* Must have computer with audio and visual capabilities.
* Must live within North Carolina
* Must have experienced health-related anxiety and/or distress in last 3 months.

Exclusion Criteria:

* Exclusion criteria will be determined by pre-screening data and medical chart reviews
* Active inpatient hospitalization
* Major cognitive impairment, marked concerns with working memory, concentration, or word finding difficulties that significantly impairs daily functioning documented in most recent clinic note or self-reported
* Recent suicide attempt(s), psychiatric hospitalization, or psychotic processing (last 3 years)
* Bipolar disorder (I or II) diagnosis, as evidenced by an ICD-10 code within the past year or revealed during subject interview
* Moderate to severe alcohol or drug abuse; as evidenced by an ICD-10 codes related to alcohol or illicit substance abuse in the medical record within the past year or revealed during subject interview.
* Severe eating disorders; as evidenced by an ICD-10 code in the medical record such as anorexia nervosa or bulimia within the past year or revealed during patient interview
* Repeated "acute" crises for example: repeated acute crises consisting of marked psychological distress that impairs function and warrants clinician intervention (e.g., occurring once a month or more frequently); this we be evaluated by the clinician screener.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katie Duckworth, Ph.D, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Among the eligible recruitment pool, direct staff member referrals were most common. The final group was comprised primarily of referrals from existing databases.
Pre-assignment Details: The most common exclusion reasons were being from outside the health system, patients/missing information or deceased prior to medical record review and non-North Carolina resident status. 55 individuals met basic study criteria, 42% cited no specific reason for declining interest or participation. 14 individuals (25%) were both eligible and interested in participating. Two people consented but did not participate. Four individuals never formally consented.
Groups:
- TeleHealth Group: The virtual group will be conducted within a secure platform such as Microsoft WebEx. Assessments (pre-, post-, mid-way) will be distributed through REDCap, a secure virtual platform, as will session handouts and forms.
  Telemental Health Sessions, Support Groups and Questionnaires: Participants will complete initial online questionnaires lasting about 25-30 minutes as well as attend weekly support group meetings online. After 4 weeks, participants will complete seven online follow-up questionnaires that should take no longer than 30 minutes and again at the end of the study.
Period: Overall Study
Arm/Group | TeleHealth Group
Started | 10
Pre-intervention Assessment | 7
Telehealth Intervention | 8
Mid-point Evaluation | 6
Completed | 6
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | TeleHealth Group
Number analyzed (Participants) | 8
Age, Continuous [Mean (Full Range); unit: years] | 26 [19 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 8
  Non-Hispanic Black | 0
  Hispanic | 0
Work/Study Location [Count of Participants; unit: Participants]
  Home | 6
  Office or School | 2
Marital Status [Count of Participants; unit: Participants]
  Single | 5
  Married | 1
  Divorced | 1
  Widowed | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Self-Efficacy in Pandemic Conditions
Description: The improvement of self-efficacy for young adult cancer survivors navigating pandemic conditions will be assessed by comparing the change in the Cancer Behaviour Inventory-Brief (CBI-B) version (a 12-item validated questionnaire used widely as a measure of self-efficacy for coping with cancer) from baseline to Visit 8. To test the change over the 8 weeks, a paired t-test (using the baseline and Visit 8 scores within the same patient) will be used; the expected difference in the CBI-B between the two scores would be no change. Score range is 1 (not at all confident) to 9 (totally confident) (minimum score of 12, maximum score of 108). Sum the scores for the 12 items with higher scores indicating greater coping efficacy.
Time Frame: At baseline up to 8 weeks
Population: Seven participants completed instruments at Baseline, 6 at 4 weeks and 8 weeks.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TeleHealth Group
Number analyzed (Participants) | 7
score on a scale
  Baseline | 86.7 [75.2 to 98.3]
  4 weeks: number analyzed (Participants) | 6
  4 weeks | 87.0 [66.1 to 107.9]
  8 weeks: number analyzed (Participants) | 6
  8 weeks | 87.8 [68.5 to 107.2]
Statistical Analysis 1: Comparison: TeleHealth Group; To test the change over the 8 weeks, a paired t-test (using the baseline and Visit 8 scores within the same patient) will be used; the expected difference in the CBI-B between the two scores would be no change. All statistical test used an alpha of 0.05; Test type: Superiority — To test the change over the 8 weeks, a paired t-test (using the baseline and Visit 8 scores within the same patient) will be used; the expected difference in the CBI-B between the two scores would be no change. All statistical test used an alpha of 0.05; p = 0.8036, t-test, 2 sided — All statistical tests were performed with a significance level of 0.05; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-7.3 to 9.0], Standard Deviation 7.8

2. Secondary Outcome: Changes in Depression and Anxiety Levels (CAS)
Description: Three instruments will provide information on baseline, Visit 8, and change over time.
  1) The Coronavirus Anxiety Scale (CAS) - 5-item mental health screener of dysfunctional anxiety associated with the coronavirus. Scoring is on a 5-point scale of 0 (not at all) to 4 (nearly every day). Minimum score (0): A score of 0 indicates that a person has not experienced any dysfunctional anxiety symptoms related to the coronavirus within the past two weeks. Maximum score (20): A score of 20 indicates the highest level of coronavirus-related anxiety, with the individual experiencing all five symptoms "nearly every day" over the past two weeks.
Time Frame: At baseline up to 8 weeks
Population: Seven participants completed instruments at Baseline, 6 at 4 weeks and 8 weeks.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TeleHealth Group
Number analyzed (Participants) | 7
score on a scale
  Baseline | 1.0 [-0.8 to 2.8]
  4 weeks: number analyzed (Participants) | 6
  4 weeks | 0.8 [-0.8 to 2.5]
  8 weeks: number analyzed (Participants) | 6
  8 weeks | 0.2 [-0.3 to 0.6]
Statistical Analysis 1: Comparison: TeleHealth Group; Test type: Superiority — Paired t-test for Coronavirus Anxiety Scale. Statistical significance using alpha of 0.05; p = 0.3632, t-test, 2 sided; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.6 to 0.3], Standard Deviation 0.4

3. Secondary Outcome: Changes in Depression and Anxiety Levels (PIL)
Description: Three instruments will provide information on baseline, Visit 8, and change over time.
  2) The Purpose in Life Test (PIL) - 20-item, 7-point Likert scale designed to measure the extent to which a respondent perceives a general sense of meaning and purpose in life using varying scale labels, scores are aggregated with a minimum score of 20 (lowest purpose) and a maximum score of 140 (highest purpose).
Time Frame: At baseline up to 8 weeks
Population: Seven participants completed instruments at Baseline, 6 at 4 weeks and 8 weeks.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TeleHealth Group
Number analyzed (Participants) | 7
score on a scale
  Baseline | 76.4 [71.2 to 81.6]
  4 weeks: number analyzed (Participants) | 6
  4 weeks | 79.3 [67.9 to 90.7]
  8 weeks: number analyzed (Participants) | 6
  8 weeks | 76.3 [61.1 to 91.5]
Statistical Analysis 1: Comparison: TeleHealth Group; Test type: Superiority — Paired t-test of Purpose in life test. Statistical significance determine with alpha of 0.05; p = 0.7918, t-test, 2 sided; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-11.3 to 9.1], Standard Deviation 9.7

4. Secondary Outcome: Changes in Depression and Anxiety Levels (MAC)
Description: Three instruments will provide information on baseline, Visit 8, and change over time.
  3) Mini-Mental Adjustments to Cancer - 29-item, 4-point Likert scale (maximum possible score of 116 and minimum possible score of 29) for rapid assessment of present coping style from 1 (Definitely Does Not Apply to Me) to 4 (Definitely Apply to Me), higher score represents higher endorsement of the adjustment response. (4). Five subscales include: Helpless-Hopeless (score range 8-32), Anxious Preoccupation (score range 8-32), Cognitive Avoidance (score range 4-16), Fighting Spirit (score range 4-16) and Fatalism (score range 5-20).
Time Frame: At baseline up to 8 weeks
Population: Seven participants completed instruments at Baseline, 6 at 4 weeks and 8 weeks.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TeleHealth Group
Number analyzed (Participants) | 7
score on a scale
  Baseline-Anxious preoccupation | 21.6 [15.2 to 28.0]
  Baseline- Cognitive avoidance | 10.1 [6.3 to 14.0]
  Baseline-Fatalism | 15.6 [12.4 to 18.7]
  Baseline- Fighting spirit | 13.4 [11.4 to 15.4]
  Baseline- Helplessness/hopelessness | 13.0 [9.4 to 16.6]
  4 weeks - Anxious preoccupation: number analyzed (Participants) | 6
  4 weeks - Anxious preoccupation | 19.2 [10.4 to 28.0]
  4 weeks - Cognitive avoidance: number analyzed (Participants) | 6
  4 weeks - Cognitive avoidance | 6.3 [4.2 to 8.5]
  4 weeks - Fatalism: number analyzed (Participants) | 6
  4 weeks - Fatalism | 15.7 [12.8 to 18.5]
  4 weeks -Fighting spirit: number analyzed (Participants) | 6
  4 weeks -Fighting spirit | 13.8 [11.8 to 15.9]
  4 weeks -Helplessness/hopelessness: number analyzed (Participants) | 6
  4 weeks -Helplessness/hopelessness | 11.5 [5.8 to 17.2]
  8 weeks- Anxious preoccupation: number analyzed (Participants) | 6
  8 weeks- Anxious preoccupation | 12.2 [6.4 to 17.9]
  8 weeks- Cognitive avoidance: number analyzed (Participants) | 6
  8 weeks- Cognitive avoidance | 7.5 [2.5 to 12.5]
  8 weeks- Fatalism: number analyzed (Participants) | 6
  8 weeks- Fatalism | 15.8 [13.1 to 18.6]
  8 weeks- Fighting spirit: number analyzed (Participants) | 6
  8 weeks- Fighting spirit | 11.0 [6.6 to 15.4]
  8 weeks- Helplessness/hopelessness: number analyzed (Participants) | 6
  8 weeks- Helplessness/hopelessness | 9.8 [7.1 to 12.6]
Statistical Analysis 1: Comparison: TeleHealth Group; Test type: Superiority — Paired t-test of The Mini-Mental Adjustment to Cancer Anxious preoccupation Subscale. Statistical significance determine with alpha of 0.05; p = 0.7711, t-test, 2 sided; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-6.2 to 4.9], Standard Deviation 5.3
Statistical Analysis 2: Comparison: TeleHealth Group; Test type: Superiority — Paired t-test of The Mini-Mental Adjustment to Cancer Cognitive avoidance Subscale. Statistical significance determine with alpha of 0.05; p = 0.0772, t-test, 2 sided; Mean Difference (Final Values) = -5.3, 95% CI 2-sided [-11.5 to 0.8], Standard Deviation 5.9
Statistical Analysis 3: Comparison: TeleHealth Group; Test type: Superiority — Paired t-test of The Mini-Mental Adjustment to Cancer Fatalism Subscale. Statistical significance determine with alpha of 0.05; p = 0.2452, t-test, 2 sided; Mean Difference (Final Values) = 3.0, 95% CI 2-sided [-2.9 to 8.9], Standard Deviation 5.6
Statistical Analysis 4: Comparison: TeleHealth Group; Test type: Superiority — Paired t-test of The Mini-Mental Adjustment to Cancer Fighting spirit Subscale. Statistical significance determine with alpha of 0.05; p = 0.6099, t-test, 2 sided; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-10.5 to 6.8], Standard Deviation 8.3
Statistical Analysis 5: Comparison: TeleHealth Group; Test type: Superiority — Paired t-test of The Mini-Mental Adjustment to Cancer Helplessness/hopelessness Subscale. Statistical significance determine with alpha of 0.05; p = 0.0913, t-test, 2 sided; Mean Difference (Final Values) = -3.0, 95% CI 2-sided [-6.7 to 0.7], Standard Deviation 3.5

ADVERSE EVENTS:
Time Frame: Deaths and adverse events were not collected.
Description: Due to the nature and scope of this study, investigators did not anticipate any adverse events would be reported by participants.
Arm/Group | TeleHealth Group
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-14): https://cdn.clinicaltrials.gov/large-docs/93/NCT04659993/Prot_SAP_001.pdf
  • Informed Consent Form (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/93/NCT04659993/ICF_000.pdf